CLINICAL TRIAL: NCT05502445
Title: Does the Nutritionist's Educational Intervention Influence Protein Intake in Hospitalized Elderly People?
Brief Title: The Nutritionist's Educational Intervention on the Protein Intake in Hospitalized Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Vanessa AC Ramis Figueira, Senior Nutritionist of Clinical Nutrition Department, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VFigueira
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Old Age; Cachexia; Dietary Habits; Sarcopenia; Protein Malnutrition; Patient Participation
Keywords: Malnutrition; Sarcopenia; Hospitalized Patients; Elderly; Patient-Centered Care; Food Intake; Protein; Nutritional Supplements
MeSH Terms: conditions — Cachexia; Feeding Behavior; Sarcopenia; Kwashiorkor; Patient Participation; Malnutrition | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: A prospective, correlational, comparative and randomized study, with hospitalized elderly over 60 years, at a private hospital.
  Patients will be randomized through a numerical sequence list, into Intervention Group (IG) or Control Group (CG). Before the nutritionist performs the first assessment, the envelope to determine which group the patient would be allocated will be selective.
  The CG will follow the flow of nutritional assessment and monitoring while the IG will receive daily visits to monitor food intake, leaflet and educational video on the importance of protein and its source foods. In both groups, a questionnaire on knowledge of protein sources and its importance will be applied, and we will calculated the 24-hour recall of a regular day and for three days of hospitalization. Patients will be assessment by Mini Nutritional Assessment-Short Form and SARC-F and will be the measurements of calf circumference and hand grip strength.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will follow the hospital's standard nutritional assessment and monitoring flow:
  * 24-hour recall: patients will be interviewed to report about one day of their usual diet.
  * Application of a questionnaire: to assess the knowledge about the importance of protein intake in the prevention of sarcopenia and functionality, and whether the participant regularly performs physical activity.
  * Energy and protein needs: estimated according to the clinical status and patient associated pathologies. The protocol of the Clinical Nutrition Service will be followed.
  * Calculation of the Body Mass Index (BMI)
  * Nutritional risk was determined using the Mini Nutritional Assessment-Short Form
  * Screening for sarcopenia: SARC-F ,Calf Circumference and Hand Grip Strength
- Intervention Group (Active Comparator): In this group, the steps below are added:
  * On the first day, the delivery of the leaflet on the importance of nutrition in the hospital environment will be added in addition to verbal guidance.
  * On the second day, an educational institutional video with duration of two minutes, will be shown with the title "Food Intake and Oral Supplement in Nutritional Rehabilitation" via tablet or mobile phone.
  * When the 24-hour recall will be collected, an assessment of food intake will be performed, mainly of foods that are sources of protein and, when they were less than 75%, strategies must be designed to increase the acceptance or indication of oral nutritional supplements (ONS).
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — In this group, the steps below are added:on the first day, the delivery of the leaflet on the importance of nutrition in the hospital environment will be added in addition to verbal guidance. On the second day, an educational institutional video with duration of two minutes, will be shown with the title "Food Intake and Oral Supplement in Nutritional Rehabilitation" via tablet or mobile phone.
  When the 24-hour recall will be collected, an assessment of food intake will be performed, mainly of foods that are sources of protein and, when they were less than 75%, strategies must be designed to increase the acceptance or indication of oral nutritional supplements.
  Arms: Intervention Group

SUMMARY:
The food intake is often compromised in the elderly, and during hospitalization, dietary restrictions may be imposed, making them more susceptible to the risk of malnutrition and sarcopenia. It is essential to make an early identification of the elderly with low intake and involve them in their self-care. The aims will be assess the influence of the nutritionist's educational action to increase protein intake in elderly patients, to analyze the knowledge on its importance in the prevention of sarcopenia and to identify the prevalence of nutritional risk. This is a field, prospective, correlational, comparative and randomized study. The elderly patients will be randomized into a Control Group and Intervention Group.

DETAILED DESCRIPTION:
The Control Group will follow the flow of nutritional assessment and monitoring while the Intervention Group will receive daily visits to monitor food intake, leaflet and educational video on the importance of protein and its source foods. In both groups, a questionnaire on knowledge of protein sources and its importance will be applied, and we will calculated the 24-hour recall of a regular day and for three days of hospitalization. Patients will be assessment by Mini Nutritional Assessment-Short Form and SARC-F and will be the measurements of calf circumference and hand grip strength.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients aged 60 years or older,
* with a prescription of oral feeding, exclusively,
* minimum period of three days.

Exclusion Criteria:

* palliative care,
* treatment for chronic renal failure,
* patients with neurological deficit and dysphagia,
* readmissions during the study,
* receiving enteral and/or parenteral nutritional therapy,
* patients in isolation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Total energy and protein needs and intakes from dietary and oral nutritional supplements during hospitalization, according to the study group | three days
  Energy and protein intakes per kg of actual body weight and per day

SECONDARY OUTCOMES:
Assessment and screening of sarcopenia risk by SARC-F questionnaire | one day (first day of assessment)
  Patients who present a result greater than or equal to 4 of this questionnaire are classified as risk of sarcopenia
Assessment of low muscle strength | one day (first day of assessment)
  The values that discriminate the altered exam are different for each age and sex. The result will be expressed as normal or low muscle strength
Assessment of low muscle mass by measuring the calf circumference | one day (first day of assessment)
  the cutoff points of 33cm for females and 34cm for males were used
Assessment and screening of nutritional risk | one day (first day of assessment)
  Assessment by Mini Nutritional Assessment-Short Form, it has the three classifications: 0-7 points: malnourished; 8 -11 points: at risk of malnutrition; or 12-14 points: well-nourished
Dietary prescription of hospitalized elderly | three days
  to evaluate the number of hospitalized elderly who remained with salt and sugar restriction in the diet, according to medical prescription
Questionnaire on previous knowledge of protein source foods and sarcopenia | one day
  The questionnaire has 9 questions related to knowledge of protein source foods and their importance on health and impact when consumption is not adequate. The last question is about physical activity, to assess how many patients follow the World Health Organization's recommendation. Was evaluated how many patients answered the questions correctly and how many practiced physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Ana P Lottenberg, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
we will available the study protocol, educational instruments applied in the intervention group (educational and video brochure) and the results of the statistical analysis
Supporting Information: Study Protocol, SAP
Time Frame: from 6 months after publication up to 2 years
Access Criteria: to obtain the study protocol and details of statistical analyses and supplementary materials, contact the author to make a request.

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Morley JE. Anorexia of ageing: a key component in the pathogenesis of both sarcopenia and cachexia. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):523-526. doi: 10.1002/jcsm.12192. Epub 2017 Apr 27. PMID 28452130
- [Background] Correia MI, Hegazi RA, Higashiguchi T, Michel JP, Reddy BR, Tappenden KA, Uyar M, Muscaritoli M. Evidence-based recommendations for addressing malnutrition in health care: an updated strategy from the feedM.E. Global Study Group. J Am Med Dir Assoc. 2014 Aug;15(8):544-50. doi: 10.1016/j.jamda.2014.05.011. Epub 2014 Jul 2. PMID 24997720
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony PS, Charlton KE, Maggio M, Tsai AC, Vellas B, Sieber CC; Mini Nutritional Assessment International Group. Frequency of malnutrition in older adults: a multinational perspective using the mini nutritional assessment. J Am Geriatr Soc. 2010 Sep;58(9):1734-8. doi: 10.1111/j.1532-5415.2010.03016.x. PMID 20863332
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Gray-Donald K, St-Arnaud-McKenzie D, Gaudreau P, Morais JA, Shatenstein B, Payette H. Protein intake protects against weight loss in healthy community-dwelling older adults. J Nutr. 2014 Mar;144(3):321-6. doi: 10.3945/jn.113.184705. Epub 2013 Dec 19. PMID 24357473
- [Background] Houston DK, Nicklas BJ, Ding J, Harris TB, Tylavsky FA, Newman AB, Lee JS, Sahyoun NR, Visser M, Kritchevsky SB; Health ABC Study. Dietary protein intake is associated with lean mass change in older, community-dwelling adults: the Health, Aging, and Body Composition (Health ABC) Study. Am J Clin Nutr. 2008 Jan;87(1):150-5. doi: 10.1093/ajcn/87.1.150. PMID 18175749
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Background] Pilgrim AL, Robinson SM, Sayer AA, Roberts HC. An overview of appetite decline in older people. Nurs Older People. 2015 Jun;27(5):29-35. doi: 10.7748/nop.27.5.29.e697. PMID 26018489
- [Background] Cox NJ, Morrison L, Ibrahim K, Robinson SM, Sayer AA, Roberts HC. New horizons in appetite and the anorexia of ageing. Age Ageing. 2020 Jul 1;49(4):526-534. doi: 10.1093/ageing/afaa014. PMID 32043144
- [Background] de van der Schueren MA, Wijnhoven HA, Kruizenga HM, Visser M. A critical appraisal of nutritional intervention studies in malnourished, community dwelling older persons. Clin Nutr. 2016 Oct;35(5):1008-14. doi: 10.1016/j.clnu.2015.12.013. Epub 2015 Dec 29. PMID 26774525
- [Background] Morley JE. Nutrition in the elderly. Curr Opin Gastroenterol. 2002 Mar;18(2):240-5. doi: 10.1097/00001574-200203000-00015. PMID 17033294
- [Background] Landi F, Picca A, Calvani R, Marzetti E. Anorexia of Aging: Assessment and Management. Clin Geriatr Med. 2017 Aug;33(3):315-323. doi: 10.1016/j.cger.2017.02.004. Epub 2017 May 20. PMID 28689565
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Effectiveness of nutritional supplementation on muscle mass in treatment of sarcopenia in old age: a systematic review. J Am Med Dir Assoc. 2013 Jan;14(1):10-7. doi: 10.1016/j.jamda.2012.08.001. Epub 2012 Sep 13. PMID 22980996
- [Background] Hope K, Ferguson M, Reidlinger DP, Agarwal E. "I don't eat when I'm sick": Older people's food and mealtime experiences in hospital. Maturitas. 2017 Mar;97:6-13. doi: 10.1016/j.maturitas.2016.12.001. Epub 2016 Dec 12. PMID 28159063
- [Background] Sieske L, Janssen G, Babel N, Westhoff TH, Wirth R, Pourhassan M. Inflammation, Appetite and Food Intake in Older Hospitalized Patients. Nutrients. 2019 Aug 22;11(9):1986. doi: 10.3390/nu11091986. PMID 31443557
- [Background] Volkert D, Beck AM, Cederholm T, Cruz-Jentoft A, Goisser S, Hooper L, Kiesswetter E, Maggio M, Raynaud-Simon A, Sieber CC, Sobotka L, van Asselt D, Wirth R, Bischoff SC. ESPEN guideline on clinical nutrition and hydration in geriatrics. Clin Nutr. 2019 Feb;38(1):10-47. doi: 10.1016/j.clnu.2018.05.024. Epub 2018 Jun 18. PMID 30005900
- [Background] Hannan-Jones M, Capra S. Developing a valid meal assessment tool for hospital patients. Appetite. 2017 Jan 1;108:68-73. doi: 10.1016/j.appet.2016.09.025. Epub 2016 Sep 22. PMID 27667562
- [Background] Roberts S, Hopper Z, Chaboyer W, Gonzalez R, Banks M, Desbrow B, Marshall AP. Engaging hospitalised patients in their nutrition care using technology: development of the NUTRI-TEC intervention. BMC Health Serv Res. 2020 Feb 27;20(1):148. doi: 10.1186/s12913-020-5017-x. PMID 32106848
- [Background] Roberts S, Desbrow B, Chaboyer W. Feasibility of a patient-centred nutrition intervention to improve oral intakes of patients at risk of pressure ulcer: a pilot randomised control trial. Scand J Caring Sci. 2016 Jun;30(2):271-80. doi: 10.1111/scs.12239. Epub 2015 Jun 2. PMID 26036929
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Barbosa-Silva TG, Bielemann RM, Gonzalez MC, Menezes AM. Prevalence of sarcopenia among community-dwelling elderly of a medium-sized South American city: results of the COMO VAI? study. J Cachexia Sarcopenia Muscle. 2016 May;7(2):136-43. doi: 10.1002/jcsm.12049. Epub 2015 Jun 9. PMID 27493867
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Introduction: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S1-S2. doi: 10.2337/dc20-Sint. No abstract available. PMID 31862741
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Background] Preston D, Nguyen TNM, Visvanathan R, Wilson A. Nutrition and the community-dwelling older person: a pilot study in general practice. Int J Evid Based Healthc. 2018 Mar;16(1):73-80. doi: 10.1097/XEB.0000000000000124. PMID 29084014
- [Background] Castro PD, Reynolds CM, Kennelly S, Geraghty AA, Finnigan K, McCullagh L, Gibney ER, Perrotta C, Corish CA. An investigation of community-dwelling older adults' opinions about their nutritional needs and risk of malnutrition; a scoping review. Clin Nutr. 2021 May;40(5):2936-2945. doi: 10.1016/j.clnu.2020.12.024. Epub 2020 Dec 23. PMID 33422348
- [Background] Avgerinou C, Bhanu C, Walters K, Croker H, Liljas A, Rea J, Bauernfreund Y, Kirby-Barr M, Hopkins J, Appleton A, Kharicha K. Exploring the Views and Dietary Practices of Older People at Risk of Malnutrition and Their Carers: A Qualitative Study. Nutrients. 2019 Jun 5;11(6):1281. doi: 10.3390/nu11061281. PMID 31195731
- [Background] Dos Santos L, Cyrino ES, Antunes M, Santos DA, Sardinha LB. Sarcopenia and physical independence in older adults: the independent and synergic role of muscle mass and muscle function. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):245-250. doi: 10.1002/jcsm.12160. Epub 2016 Nov 8. PMID 27897417
- [Background] Diz JB, Leopoldino AA, Moreira BS, Henschke N, Dias RC, Pereira LS, Oliveira VC. Prevalence of sarcopenia in older Brazilians: A systematic review and meta-analysis. Geriatr Gerontol Int. 2017 Jan;17(1):5-16. doi: 10.1111/ggi.12720. Epub 2016 Jan 22. PMID 26799062
- [Background] Tieland M, Borgonjen-Van den Berg KJ, Van Loon LJ, de Groot LC. Dietary Protein Intake in Dutch Elderly People: A Focus on Protein Sources. Nutrients. 2015 Nov 25;7(12):9697-706. doi: 10.3390/nu7125496. PMID 26610565
- [Background] Ten Haaf DSM, van Dongen EJI, Nuijten MAH, Eijsvogels TMH, de Groot LCPGM, Hopman MTE. Protein Intake and Distribution in Relation to Physical Functioning and Quality of Life in Community-Dwelling Elderly People: Acknowledging the Role of Physical Activity. Nutrients. 2018 Apr 19;10(4):506. doi: 10.3390/nu10040506. PMID 29671766
- [Background] Weijzen MEG, Kouw IWK, Geerlings P, Verdijk LB, van Loon LJC. During Hospitalization, Older Patients at Risk for Malnutrition Consume <0.65 Grams of Protein per Kilogram Body Weight per Day. Nutr Clin Pract. 2020 Aug;35(4):655-663. doi: 10.1002/ncp.10542. Epub 2020 Jun 24. PMID 32578906
- [Background] Ingadottir AR, Beck AM, Baldwin C, Weekes CE, Geirsdottir OG, Ramel A, Gislason T, Gunnarsdottir I. Association of energy and protein intakes with length of stay, readmission and mortality in hospitalised patients with chronic obstructive pulmonary disease. Br J Nutr. 2018 Mar;119(5):543-551. doi: 10.1017/S0007114517003919. PMID 29508694
- [Background] Dijxhoorn DN, IJmker-Hemink VE, Wanten GJA, van den Berg MGA. Strategies to increase protein intake at mealtimes through a novel high-frequency food service in hospitalized patients. Eur J Clin Nutr. 2019 Jun;73(6):910-916. doi: 10.1038/s41430-018-0288-6. Epub 2018 Aug 22. PMID 30135550
- [Background] Vasse E, Beelen J, de Roos NM, Janssen N, de Groot LC. Protein intake in hospitalized older people with and without increased risk of malnutrition. Eur J Clin Nutr. 2018 Jun;72(6):917-919. doi: 10.1038/s41430-018-0171-5. Epub 2018 May 15. PMID 29760481
- See also: Vigitel Brazil 2019:surveillance of risk and protect.factors for chronic dis.by telephone survey: estimates of frequency and sociodemographic distribution of risk and protect.factors for chronic dis.in the capitals in 2019 — https://www.saude.gov.br/svs
- See also: World Health Organization. (2020). WHO guidelines on physical activity and sedentary behaviour: at a glance. World Health Organization. https://apps.who.int/iris/handle/10665/337001 — https://apps.who.int/iris/handle/10665/337001
- See also: World Health Organization. (2002, april). Active Ageing - A Policy Framework. A contribution of the World Health Organization to the Second United Nations World Assembly on Ageing. p.4. [Accessed on August 22, 2020] — https://extranet.who.int/agefriendlyworld/wp-content/uploads/2014/06/WHO-Active-Ageing-Framework.pdf
- See also: Gonçalves, TJM e col. BRASPEN. Brazilian Society of Parenteral and Enteral Nutrition. Guideline on nutrition therapy in aging. J 2019; 34 (Supl 3):2-58) — https://www.braspen.org/diretrizes